CLINICAL TRIAL: NCT06308913
Title: Pilot Study of INCB081776 Together With Palliative Radiation and Anti-PD-1 Checkpoint Blockade With Pembrolizumab in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Pembrolizumab, INCB081776, and Radiation Therapy for Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1722; UW23121 (Other: UWCCC); A534260 (Other: UW Madison); Protocol Version 6/3/2025 (Other: UW Madison); P50CA278595 (NIH)
Record Dates: First submitted 2024-03-05; First posted 2024-03-13 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: metastatic
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INCB081776/Pembrolizumab and RT for HNSCC (Experimental): Cycle 1 of this clinical trial is 56 days in duration to allow for the systematic addition of each agent to the combination regimen. For cycle 2 and all subsequent cycles, the treatment cycle will be 21 days in length.
  Interventions: Drug: INCB081776; Drug: Pembrolizumab; Radiation: Palliative RT

INTERVENTIONS:
Drug: INCB081776 — INCB081776 will be given orally on a daily basis. The highest safe/tolerable dose and schedule will be established by the ongoing phase 1 clinical trial of INCB081776 plus INCBMGA00012 (NCT03522142), which is 120 mg daily.
Drug: Pembrolizumab — Immune checkpoint blockade with anti-PD-1 (Pembrolizumab) will be given as 200 mg IV on cycle 1 day 15 and cycle 1 day 36. Starting from cycle 2, pembrolizumab will be given on day 1 on each subsequent cycle.
Radiation: Palliative RT — Palliative RT will be given as either 24 Gy in 3 fractions (8 Gy per fraction) or 20 Gy in 5 fractions (4 Gy per fraction). The palliative radiation therapy dose will be determined based on the clinical judgment of the treating radiation oncology physician. Palliative RT must be completed between cycle 1 day 29 to cycle 1 day 33. After completion of palliative radiation therapy, patients will continue with additional cycles of INCB081776 and pembrolizumab until disease progression, intolerance to the combination regimen, or patient withdrawal.

SUMMARY:
This study is evaluating INCB081776 when given in combination with the checkpoint inhibitor pembrolizumab and palliative radiation therapy in patients with metastatic or recurrent metastatic or recurrent head and neck squamous cell carcinoma (HNSCC). 12 participants will be enrolled and can expect to be on study for up to 12 months.

DETAILED DESCRIPTION:
Primary Objective

• To evaluate the safety and tolerability of INCB081776 in combination with pembrolizumab and standard palliative radiation therapy in subjects with recurrent/metastatic squamous cell carcinoma of the head and neck.

Secondary Objectives

• To determine the preliminary efficacy of INCB081776 in combination with pembrolizumab plus palliative radiation therapy in subjects with recurrent/metastatic squamous cell carcinoma of the head and neck. The irradiated lesion (lesion A) will not be included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologic or cytologic evidence of head and neck squamous cell carcinoma (HNSCC) that is metastatic or recurrent and therefore considered incurable. Cutaneous skin squamous cell carcinomas located in the head and neck region are eligible after discussion with the Sponsor-Investigator.
* Measurable disease that are considered non-amenable to surgery or other curative treatments or procedures, with at least 1 target lesion available for evaluation.

  * The preference is for measurable disease to be selected from a site that has not received any prior radiation or locoregional therapy. However, if a tumor lesion is situated in a previously irradiated area, or in an area subjected to other prior locoregional therapy, the lesion should demonstrate disease progression after the prior treatment.
* Prior cancer treatment must be completed at least 14 days prior to enrollment (for chemotherapy, targeted small molecular therapy, or radiation therapy. Prior treatment with a monoclonal antibody must be completed at least 28 days prior to enrollment. Participants must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to ≤ Grade 1 or baseline.
* Participants must have two "index" tumors that meet the following criteria:

  * Index tumor A (lesion to receive palliative radiation therapy):

    * is deemed by the treating radiation oncologist to potentially benefit from palliative radiation
    * is at least 1 cm in longest dimension for lesions not located in the bone, if radiating bone, presence of a bone lesion is sufficient.
  * Index tumor B (lesion to undergo biopsy):

    * Is deemed by the treating physician to be amenable to biopsy
    * Is at least 1 cm in longest dimension.
    * Participants must be willing to provide at least 2 research biopsies (up to 3 research biopsies) during the conduct of the study.
    * Note: If a subject is scheduled to have a baseline or on-study tumor biopsy, and the investigator believes that the tumor tissue cannot be obtained safely, then the biopsy may be omitted with approval by the Sponsor-Investigator. The participant may be replaced in order to enroll sufficient number of subjects for biomarker evaluation.
    * Note: Care should be taken to biopsy the same lesions for research samples. The preference is for the same lesion to be biopsied at all time points. If a lesion is no longer amenable for a research biopsy (for examples: due to a decrease in size, becomes inaccessible, is not safe/feasible for a biopsy), then an alternative lesion may be utilized with approval by the Sponsor-Investigator. Index tumor B (lesion to undergo biopsy) must not have received palliative radiation therapy during the study.
* Participants must be willing to provide at least 2 collections of fresh research biopsies (up to 3 fresh research biopsies) during the conduct of this study.

  * Research biopsy #1 (baseline, mandatory). Archival tissue obtained since completion of last therapy may be used.
  * Research biopsy #2 (cycle 1 days 9-14, after treatment with INCB081776 but prior to pembrolizumab, mandatory)
  * Research biopsy #3 (cycle 1 day 37-56, after treatment with INCB081776, pembrolizumab and palliative RT). For participants who had baseline archival tissue collected (no baseline research biopsy was obtained), this fresh core biopsy is mandatory. For participants who underwent a fresh core research biopsy at baseline, this biopsy is optional.
  * Note: If a participant is scheduled to have an on-study tumor biopsy, and the investigator believes that the tumor tissue cannot be obtained safely, then the biopsy may be omitted after discussion with the Sponsor-Investigator. The participant may be replaced in order to enroll sufficient number of subjects for biomarker evaluation.
  * Note: Care should be taken to biopsy the same lesion for the on-treatment samples

Exclusion Criteria:

* Subjects with significant intercurrent illnesses per physician discretion.
* Subjects with a diagnosed auto-immune disease requiring systemic treatment with immunosuppressants.
* Subjects with known genetic conditions causing pre-disposition to RT toxicity (i.e: Li-Fraumeni, ATM deficiency, active scleroderma, etc.).
* Subjects with known retinal or ophthalmologic disorders or conditions. Subjects with macular degeneration, proliferative diabetic retinopathy or diabetic retinopathy with macular edema, retinal vein occlusions, uveitis, central serous retinopathy, leukemic retinopathy, inherited retinal degenerations, known family history of inherited retinal degenerations, and subjects at risk for angle closure glaucoma from pupillary dilation are ineligible. Subjects with other clinically significant abnormalities identified during ophthalmic screening examinations that may confound ocular monitoring are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Participants will be followed for 30 days (+/- 7 days) after the last dose of treatment (up to 12 months on study)
  Frequency of AEs through physical examinations, by evaluating changes in vital signs, through clinical laboratory blood sample evaluations.
Duration of Adverse Events | Participants will be followed for 30 days (+/- 7 days) after the last dose of treatment (up to 12 months on study)
  Duration of AEs through physical examinations, by evaluating changes in vital signs, through clinical laboratory blood sample evaluations.
Severity of Adverse Events | Participants will be followed for 30 days (+/- 7 days) after the last dose of treatment (up to 12 months on study)
  Severity of AEs through physical examinations, by evaluating changes in vital signs, through clinical laboratory blood sample evaluations. Severity will be reported by Grade between 1 (mild) and 5 (death).

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to 12 months
  Defined as the percentage of participants having CR or PR per RECIST 1.1. The irradiated lesion (lesion A) will not be included in the analysis.
Disease control rate (DCR) | up to 12 months
  Defined as the percentage of participants having complete response (CR), partial response (PR), or stable disease (SD) per RECIST 1.1.
Duration of response (DoR) | up to 12 months
  Defined as the time from earliest date of response until the earliest date of disease progression or death per RECIST 1.1 due to any cause, if occurring sooner than progression.

CONTACTS AND LOCATIONS:
Overall Officials: Justine Bruce, MD, Principal Investigator — University of Wisconsin, Madison; Deric Wheeler, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No